CLINICAL TRIAL: NCT01011868
Title: A Phase IIb, Randomized, Double-blind, Placebo-controlled, Parallel Group, Safety and Efficacy Study of BI 10773 (10 mg and 25 mg) Administered Orally, Once Daily Over 78 Weeks in Type 2 Diabetic Patients Receiving Treatment With Basal Insulin (Glargine, Detemir, or NPH Insulin Only) With or Without Concomitant Metformin and/or Sulfonylurea Therapy and Insufficient Glycemic Control
Brief Title: Efficacy and Safety of BI 10773 in Combination With Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.33; 2009-013668-38 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (3):
- BI 10773 low dose (Experimental): Patients receive BI 10773 low dose daily
  Interventions: Drug: BI 10773 low dose
- BI 10773 high dose (Experimental): Patients receive BI 10773 high dose daily
  Interventions: Drug: BI 10773 placebo; Drug: BI 10773 high dose
- placebo (Placebo Comparator): Patients receive placebo to match BI 10773 daily
  Interventions: Drug: BI 10773 placebo

INTERVENTIONS:
Drug: BI 10773 placebo — BI 10773 placebo
  Arms: BI 10773 high dose
Drug: BI 10773 low dose — BI 10773 low dose
  Arms: BI 10773 low dose
Drug: BI 10773 high dose — BI 10773 high dose
  Arms: BI 10773 high dose
Drug: BI 10773 placebo — BI 10773 placebo
  Arms: placebo

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of BI 10773 at two different doses compared to placebo during long term treatment (78 weeks) in combination with basal insulin in patients with type 2 diabetes mellitus with insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation
2. Male and female patients with a diagnosis of Type 2 Diabetes Mellitus treated with a stable dose of basal insulin with or without concomitant metformin and / or sulfonylurea.
3. Glycosylated hemoglobin A1c (Type A, subtype 1c) of >7.0% and < or = 10% at Visit 1 (screening)
4. Suitability for trial participation according to investigator's judgment (evaluating all alternative treatment options and in consideration of the patient completing the study)
5. Age > or =18 years at Visit 1 (screening)
6. BMI < or = 45 kg/m2 (Body Mass Index) at Visit 1 (screening)

Exclusion criteria:

1. Patients with poorly controlled hyperglycemia
2. Frequent (at the discretion of the investigator) episodes of hypoglycemic events on basal insulin therapy
3. MI, stroke, or TIA within 3 months prior to obtaining informed consent
4. Impaired hepatic or renal function; gastric surgery; cancer within the last 5 years; blood dyscrasias

6. Treatment with other anti-diabetics, anti-obesity medications, steroids or thyroid hormones, participation in another trial with an investigational drug 7. Pre-menopausal women on insufficient birth control 8. Alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (99):
- United States (56):
  - 1245.33.01014 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1245.33.01047 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1245.33.01060 Boehringer Ingelheim Investigational Site, Fresno, California
  - 1245.33.01013 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1245.33.01008 Boehringer Ingelheim Investigational Site, Los Gatos, California
  - 1245.33.01019 Boehringer Ingelheim Investigational Site, National City, California
  - 1245.33.01055 Boehringer Ingelheim Investigational Site, Paramount, California
  - 1245.33.01012 Boehringer Ingelheim Investigational Site, Santa Ana, California
  - 1245.33.01054 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1245.33.01046 Boehringer Ingelheim Investigational Site, Bradednton, Florida
  - 1245.33.01050 Boehringer Ingelheim Investigational Site, Brooksville, Florida
  - 1245.33.01059 Boehringer Ingelheim Investigational Site, Chiefland, Florida
  - 1245.33.01028 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1245.33.01029 Boehringer Ingelheim Investigational Site, Fleming Island, Florida
  - 1245.33.01048 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1245.33.01033 Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - 1245.33.01027 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1245.33.01040 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1245.33.01062 Boehringer Ingelheim Investigational Site, Lawrenceville, Georgia
  - 1245.33.01020 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1245.33.01044 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1245.33.01024 Boehringer Ingelheim Investigational Site, Des Moines, Iowa
  - 1245.33.01022 Boehringer Ingelheim Investigational Site, Saint Louis, Maryland
  - 1245.33.01056 Boehringer Ingelheim Investigational Site, Olive Branch, Mississippi
  - 1245.33.01032 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1245.33.01017 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1245.33.01043 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1245.33.01051 Boehringer Ingelheim Investigational Site, New Hartford, New York
  - 1245.33.01007 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 1245.33.01003 Boehringer Ingelheim Investigational Site, Jacksonville, North Carolina
  - 1245.33.01016 Boehringer Ingelheim Investigational Site, Salisbury, North Carolina
  - 1245.33.01005 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 1245.33.01038 Boehringer Ingelheim Investigational Site, Wilmington, North Carolina
  - 1245.33.01026 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1245.33.01025 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.33.01001 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1245.33.01031 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1245.33.01045 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 1245.33.01018 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 1245.33.01041 Boehringer Ingelheim Investigational Site, Carlisle, Pennsylvania
  - 1245.33.01042 Boehringer Ingelheim Investigational Site, Landsdale, Pennsylvania
  - 1245.33.01004 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1245.33.01036 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 1245.33.01035 Boehringer Ingelheim Investigational Site, Seneca, South Carolina
  - 1245.33.01058 Boehringer Ingelheim Investigational Site, Kingsport, Tennessee
  - 1245.33.01037 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1245.33.01023 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.33.01030 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.33.01006 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.33.01011 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.33.01002 Boehringer Ingelheim Investigational Site, Sugar Land, Texas
  - 1245.33.01049 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1245.33.01015 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 1245.33.01009 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1245.33.01010 Boehringer Ingelheim Investigational Site, Federal Way, Washington
  - 1245.33.01061 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Denmark (8):
  - 1245.33.45006 Boehringer Ingelheim Investigational Site, Aalborg
  - 1245.33.45001 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1245.33.45011 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1245.33.45013 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1245.33.45004 Boehringer Ingelheim Investigational Site, Gentofte Municipality
  - 1245.33.45008 Boehringer Ingelheim Investigational Site, Hillerød
  - 1245.33.45002 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1245.33.45003 Boehringer Ingelheim Investigational Site, København NV
- France (9):
  - 1245.33.3301A Boehringer Ingelheim Investigational Site, Bondy
  - 1245.33.3302A Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - 1245.33.3305A Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.33.3306A Boehringer Ingelheim Investigational Site, Marseille
  - 1245.33.3308A Boehringer Ingelheim Investigational Site, Montbrison
  - 1245.33.3309A Boehringer Ingelheim Investigational Site, Nanterre
  - 1245.33.3310A Boehringer Ingelheim Investigational Site, Nantes
  - 1245.33.3304A Boehringer Ingelheim Investigational Site, Narbonne
  - 1245.33.3303A Boehringer Ingelheim Investigational Site, Saint-Mandé
- Ireland (3):
  - 1245.33.35302 Boehringer Ingelheim Investigational Site, Dublin
  - 1245.33.35303 Boehringer Ingelheim Investigational Site, Dublin
  - 1245.33.35304 Boehringer Ingelheim Investigational Site, Dublin
- Portugal (5):
  - 1245.33.35104 Boehringer Ingelheim Investigational Site, Aveiro
  - 1245.33.35101 Boehringer Ingelheim Investigational Site, Coimbra
  - 1245.33.35102 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.33.35106 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.33.35107 Boehringer Ingelheim Investigational Site, Lisbon
- South Korea (8):
  - 1245.33.82008 Boehringer Ingelheim Investigational Site, Daejeon
  - 1245.33.82007 Boehringer Ingelheim Investigational Site, Gwangju
  - 1245.33.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.33.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.33.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.33.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.33.82006 Boehringer Ingelheim Investigational Site, Wŏnju
  - 1245.33.82002 Boehringer Ingelheim Investigational Site, Yangsan
- United Kingdom (10):
  - 1245.33.44001 Boehringer Ingelheim Investigational Site, Bath
  - 1245.33.44003 Boehringer Ingelheim Investigational Site, Birmingham
  - 1245.33.44006 Boehringer Ingelheim Investigational Site, Blackburn
  - 1245.33.44005 Boehringer Ingelheim Investigational Site, Dorking
  - 1245.33.44009 Boehringer Ingelheim Investigational Site, Headington
  - 1245.33.44008 Boehringer Ingelheim Investigational Site, Leicester
  - 1245.33.44004 Boehringer Ingelheim Investigational Site, Liverpool
  - 1245.33.44007 Boehringer Ingelheim Investigational Site, Wembley
  - 1245.33.44002 Boehringer Ingelheim Investigational Site, Whitstable
  - 1245.33.44010 Boehringer Ingelheim Investigational Site, Wymondham

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral Placebo
- Empagliflozin 10 mg: Empagliflozin 10 mg orally once daily
- Empagliflozin 25 mg: Empagliflozin 25 mg orally once daily
Period: After Week 18 Follow-up
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 170 | 169 | 155
Completed | 147 | 153 | 129
Not Completed | 23 | 16 | 26
Not completed — Adverse Event | 8 | 6 | 13
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Lost to Follow-up | 5 | 3 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 0
Not completed — Other reason not defined above | 2 | 3 | 12
Period: After Week 78 Follow-up
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 170 | 169 | 155
Completed | 118 | 131 | 111
Not Completed | 52 | 38 | 44
Not completed — Adverse Event | 14 | 18 | 21
Not completed — Lack of Efficacy | 4 | 0 | 0
Not completed — Protocol Violation | 9 | 1 | 2
Not completed — Lost to Follow-up | 11 | 6 | 4
Not completed — Withdrawal by Subject | 9 | 8 | 1
Not completed — Other reason not defined above | 5 | 5 | 16

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) - including all randomized and treated patients who had a baseline HbA1c value. Treatment assignment as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 170 | 169 | 155 | 494
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.4) | 58.6 (9.8) | 59.9 (10.5) | 58.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 76 | 62 | 218
  Male | 90 | 93 | 93 | 276

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) After 18 Weeks of Treatment
Description: Change from baseline in Glycosylated haemoglobin A1c (HbA1c) after 18 weeks of treatment
Time Frame: Baseline and 18 weeks
Population: FAS18-completers-included FAS patients not prematurely discontinue prior to Week 18, completed required minimum treatment duration, and had an on treatment HbA1c value within Week 18 time window. Values after start of antidiabetic rescue therapy were set to missing and last observation carried forward (LOCF-18) was used for imputation.
  (LOCF-18)
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 125 | 132 | 117
percentage of HbA1c | 0.03 (0.07) | -0.58 (0.07) | -0.75 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; The null and alternative hypotheses to be tested: * H0,1: No difference in change from baseline to Week 18 in HbA1c between empagliflozin 10 mg and placebo * H1,1: A difference in change from baseline to Week 18 in HbA1c between empagliflozin 10 mg and placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hypotheses were tested at significance level of 0.025, which is half of overall alpha of 0.05, split equally between 2 treatment comparisons. This maintained the overall type-I (alpha) at 5%. There was no a priori assumption on testing order; ANCOVA that included treatment group and geographic region as fixed effects along with baseline HbA1c as covariate; Adjusted mean difference = -0.56, 97.5% CI 2-sided [-0.78 to -0.33], Standard Error of Mean 0.10 — The primary analysis consisted of the pair-wise comparisons between each dose of empagliflozin versus placebo using the adjusted means from the model
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; The null and alternative hypotheses to be tested: * H0,2: No difference in change from baseline to Week 18 in HbA1c between empagliflozin 25 mg and placebo * H1,2: A difference in change from baseline to Week 18 in HbA1c between empagliflozin 25 mg and placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA that included treatment group and geographic region as fixed effects along with baseline HbA1c as covariate; Adjusted mean difference = -0.70, 97.5% CI 2-sided [-0.93 to -0.47], Standard Error of Mean 0.10 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Occurrence of Relative Efficacy Response (HbA1c Lowering by at Least 0.5%) After 18, 54 and 78 Weeks of Treatment
Description: Patients that had a reduction in HbA1c of at least 0.5% from baseline to 18, 54 and 78 weeks of treatment
Time Frame: Baseline and 18, 54 and 78 weeks
Population: FAS with non-completers considered failure (NCF)
Measure: Number; unit: participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 170 | 169 | 155
participants
  18 weeks | 27 | 85 | 73
  54 weeks | 30 | 72 | 69
  78 weeks | 27 | 59 | 61
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Empagliflozin 10 mg vs Placebo at 18 weeks; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 5.518, 95% CI 2-sided [3.262 to 9.334]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Empagliflozin 25 mg vs Placebo at 18 weeks; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 4.883, 95% CI 2-sided [2.859 to 8.338]
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 10 mg; Empagliflozin 10 mg vs Placebo at 54 weeks; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 3.471, 95% CI 2-sided [2.077 to 5.802]
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Empagliflozin 25 mg vs Placebo at 54 weeks; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 3.825, 95% CI 2-sided [2.268 to 6.451]
Statistical Analysis 5: Comparison: Placebo vs Empagliflozin 10 mg; Empagliflozin 10 mg vs Placebo at 78 weeks; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 2.802, 95% CI 2-sided [1.639 to 4.789]
Statistical Analysis 6: Comparison: Placebo vs Empagliflozin 25 mg; Empagliflozin 25 mg vs Placebo at 78 weeks; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 3.527, 95% CI 2-sided [2.051 to 6.066]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 18, 54 and 78 Weeks of Treatment
Description: Change from baseline in fasting plasma glucose (FPG) after 18, 54 and 78 weeks of treatment
Time Frame: Baseline, 18, 54 and 78 weeks
Population: FAS observed cases (OC)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 135 | 138 | 120
mg/dL
  week 18 Change from BL | 9.81 (5.48) | -14.79 (3.93) | -27.03 (3.92)
  week 54 Change from BL (N=103,111,99) | 0.91 (5.08) | -9.59 (4.69) | -23.75 (4.62)
  week 78 Change from BL (N=92,104,92) | -5.53 (4.95) | -7.75 (4.66) | -21.62 (5.13)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 18 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Model includes, baseline FPG, baseline HbA1c as covariates, geographic region, treatment, visit and visit by treatment interaction as fixed effects; Adjusted mean difference = -28.40, 95% CI 2-sided [-37.54 to -19.27], Standard Error of Mean 4.65
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 18 - Empagliflozin 25 mg vs Placebo at 18 weeks; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -34.21, 95% CI 2-sided [-43.67 to -24.76], Standard Error of Mean 4.81
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 54 - Empagliflozin 10 mg vs Placebo at 18 weeks; Test type: Superiority or Other; p = 0.0328, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -10.75, 95% CI 2-sided [-20.62 to -0.89], Standard Error of Mean 5.02
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 54 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -19.16, 95% CI 2-sided [-29.31 to -9.01], Standard Error of Mean 5.16
Statistical Analysis 5: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 78 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p = 0.3216, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -5.03, 95% CI 2-sided [-15.01 to 4.94], Standard Error of Mean 5.07
Statistical Analysis 6: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 78 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.0229, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -11.95, 95% CI 2-sided [-22.24 to -1.67], Standard Error of Mean 5.23

4. Secondary Outcome: Percent Change From Baseline in Fasting Plasma Glucose (FPG) After 18, 54 and 78 Weeks of Treatment
Description: Percent change from baseline in fasting plasma glucose (FPG) after 18, 54 and 78 weeks of treatment
Time Frame: Baseline, 18, 54 and 78 weeks
Population: FAS (OC)
Measure: Mean (Standard Error); unit: percentage of Change from BL in FPG
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 135 | 138 | 120
percentage of Change from BL in FPG
  week 18 % CHG | 19.02 (6.32) | -2.80 (3.17) | -13.43 (2.39)
  week 54 % CHG (N=103,111,99) | 9.67 (5.58) | 0.67 (4.05) | -11.59 (3.04)
  week 78 % CHG (N=92,104,92) | 4.75 (5.67) | 2.43 (4.18) | -9.52 (3.40)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 18 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -25.12, 95% CI 2-sided [-35.38 to -14.86], Standard Error of Mean 5.22
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 18 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -31.01, 95% CI 2-sided [-41.62 to -20.39]
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 54 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p < 0.0484, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -10.20, 95% CI 2-sided [-20.33 to -0.07], Standard Error of Mean 5.15
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 54 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -19.42, 95% CI 2-sided [-29.84 to -8.99], Standard Error of Mean 5.30
Statistical Analysis 5: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 78 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p = 0.3517, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -4.73, 95% CI [-14.71 to 5.25], Standard Error of Mean 5.07
Statistical Analysis 6: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 78 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.0185, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -12.39, 95% CI 2-sided [-22.69 to -2.10], Standard Error of Mean 5.23

5. Secondary Outcome: Change From Baseline in Basal Insulin Dose/Day After 54 and 78 Weeks of Treatment
Description: Change from baseline in basal insulin dose/day after 54 and 78 weeks of treatment
Time Frame: Baseline, 54 and 78 weeks
Population: FAS (OC-78) for week 54 FAS78-completers (LOCF-78) for week 78 - Values after start of antidiabetic rescue therapy except changes in basal insulin dose were set to missing and last observation carried forward (LOCF) was used for imputation of missing values
Measure: Mean (Standard Error); unit: IU
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 112 | 127 | 110
IU
  week 54 (N=112,122,104) | 5.39 (1.60) | -1.20 (1.40) | -1.12 (1.27)
  week 78 | 4.79 (2.06) | -0.70 (1.85) | -0.39 (1.06)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Empagliflozin versus Placebo 10 mg at 54 weeks; Test type: Superiority or Other; p = 0.0213, Mixed Models Analysis; Adjusted mean difference = -5.58, 95% CI 2-sided [-10.32 to -0.84], Standard Error of Mean 2.40 — Week 54 model includes, baseline basal insulin, baseline HbA1c as linear covariate(s), geographical region, treatment, visit and visit by treatment interaction as fixed effects
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Empagliflozin versus Placebo 25 mg at 54 weeks; Test type: Superiority or Other; p = 0.0237, Mixed Models Analysis; Adjusted mean difference = -5.69, 95% CI 2-sided [-10.62 to -0.77], Standard Error of Mean 2.49 — Week 54 model includes, baseline basal insulin, baseline HbA1c as linear covariate(s), geographical region, treatment, visit and visit by treatment interaction as fixed effect(s)
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 10 mg; Empagliflozin versus Placebo 10 mg at 78 weeks H0,1a: No difference in change from baseline to Week 78 in basal insulin dose between Empagliflozin 10 mg and placebo H1,1a: A difference in change from baseline to Week 78 in basal insulin dose between Empagliflozin 10 mg and placebo; Test type: Superiority or Other; p = 0.0024, ANCOVA — Hierarchical testing approach was applied to Empagliflozin 10 mg vs Placebo. If null hypothesis is rejected for the primary endpoint, at 0.025 (2-sided), testing of the key secondary endpoints continued in a hierarchical fashion for the same dose; Model for Week 78 includes baseline basal insulin, baseline HbA1c as linear covariate(s) and geographical region, treatment as fixed effect(s); Adjusted mean difference = -6.66, 97.5% CI 2-sided [-11.56 to -1.77], Standard Error of Mean 2.18
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Empagliflozin versus Placebo 25 mg at 78 weeks H0,1a: No difference in change from baseline to Week 78 in basal insulin dose between Empagliflozin 25 mg and placebo H1,1a: A difference in change from baseline to Week 78 in basal insulin dose between Empagliflozin 25 mg and placebo; Test type: Superiority or Other; p = 0.0090, ANCOVA — Hierarchical testing approach was applied to Empagliflozin 25 mg vs Placebo. If null hypothesis is rejected for the primary endpoint, at 0.025 (2-sided), testing of the key secondary endpoints continued in a hierarchical fashion for the same dose; [statistical method as in outcome 5, analysis 3]; Adjusted mean difference = -5.92, 97.5% CI 2-sided [-11.00 to -0.85], Standard Error of Mean 2.25

6. Secondary Outcome: Change From Baseline in Body Weight After 18, 54 and 78 Weeks of Treatment
Description: Change from baseline in body weight after 18, 54 and 78 weeks of treatment
Time Frame: Baseline, 18, 54, 78 weeks
Population: FAS (OC)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 141 | 148 | 125
kg
  18 weeks | -0.04 (0.21) | -2.06 (0.22) | -0.91 (1.27)
  54 weeks (N=114,120,106) | -0.52 (0.32) | -2.28 (0.33) | -2.23 (0.35)
  78 weeks (N=100,113,96) | 1.12 (1.28) | -2.61 (0.31) | -1.99 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 18 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p = 0.0320, Mixed Models Analysis; Adjusted mean difference = -2.04, 95% CI 2-sided [-3.90 to -0.18], Standard Error of Mean 0.95 — Model includes baseline weight, baseline HbA1c as linear covariates, geographical region, treatment, visit and visit by treatment interaction as fixed effects
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 18 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.3818, Mixed Models Analysis; Adjusted mean difference = -0.87, 95% CI 2-sided [-2.81 to 1.08], Standard Error of Mean 0.99 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 54 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted mean difference = -1.97, 95% CI 2-sided [-2.89 to -1.05], Standard Error of Mean 0.47 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 54 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted mean difference = -2.17, 95% CI 2-sided [-3.13 to -1.22], Standard Error of Mean 0.49 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 78 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; Adjusted mean difference = -3.63, 95% CI 2-sided [-5.81 to -1.45], Standard Error of Mean 1.10 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 78 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis; Model includes, baseline weight, baseline HbA1c as covariates, geographic region, treatment, visit and visit by treatment interaction as fixed effects; Adjusted mean difference = -3.12, 95% CI 2-sided [-5.39 to -0.85], Standard Error of Mean 1.15 — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in Body Weight at Follow-up
Description: Change from baseline in body weight at follow up (82 weeks)
Time Frame: Baseline and 82 weeks
Population: FAS-FU (OR)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 111 | 119 | 112
kg
  Follow-up | 90.56 (25.87) | 90.44 (19.35) | 93.98 (20.87)
  Follow-up change from baseline | 0.92 (12.20) | -2.02 (4.04) | -1.05 (3.96)
  Change from last value on treatment N=111,118,109 | -0.23 (16.84) | 0.62 (2.11) | 1.34 (1.90)

8. Secondary Outcome: Change From Baseline in HbA1c After 54 and 78 Weeks of Treatment
Description: Change from baseline in HbA1c after 54 and 78 weeks of treatment
Time Frame: Baseline, 54 and 78 weeks
Population: Week 54 - FAS (OC-78) Week 78 - FAS78-completers (LOCF-78)
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 113 | 127 | 110
percentage of HbA1c
  Week 54 (N=113,121,107) | -0.06 (0.08) | -0.59 (0.08) | -0.84 (0.09)
  Week 78 (N=112,127,110) | -0.05 (0.10) | -0.51 (0.09) | -0.68 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 54 - Empagliflozin 10 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted mean difference = -0.47, 95% CI 2-sided [-0.68 to -0.26], Standard Error of Mean 0.11 — Model includes baseline HbA1c as linear covariate(s), geographical region, treatment, visit and visit by treatment interaction as fixed effect(s)
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 54 - Empagliflozin 25 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted mean difference = -0.74, 95% CI 2-sided [-0.95 to -0.52], Standard Error of Mean 0.11 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 10 mg; Change from BL at week 78 - Empagliflozin 10 mg vs Placebo H0,1b: The change from baseline to Week 78 in HbA1c between empagliflozin 10 mg and placebo ≥0.3% H1,1b: The change from baseline to Week 78 in HbA1c between empagliflozin 10 mg and placebo <0.3%; Test type: Non-Inferiority or Equivalence — For non-inferiority, a one-sided test at the significance level of 0.0125 was performed using a chosen margin of 0.3% difference between each dose of empagliflozin and placebo. If the non-inferiority of empagliflozin to placebo with respect to change from baseline in HbA1c after 78 weeks of treatment could be concluded for a specific dose, subsequent testing of superiority was performed at the significance level of 0.025 for the relevant empagliflozin dose versus placebo comparison; p = 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 3]; Adjusted mean difference = -0.46, 97.5% CI 2-sided [-0.73 to -0.19], Standard Error of Mean 0.12 — Model includes baseline HbA1c as linear covariate(s), geographical region, treatment as fixed effect(s)
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Change from BL at week 78 - Empagliflozin 25 mg vs Placebo H0,1b: The change from baseline to Week 78 in HbA1c between empagliflozin 25 mg and placebo ≥0.3% H1,1b: The change from baseline to Week 78 in HbA1c between empagliflozin 25 mg and placebo <0.3%; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 3]; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 4]; Adjusted mean difference = -0.62, 97.5% CI 2-sided [-0.90 to -0.34], Standard Error of Mean 0.12 — Model includes baseline HbA1c as linear covariate(s), geographical region, treatment as fixed effect(s)

9. Other Pre Specified Outcome: Confirmed Hypoglycemic Events
Description: Confirmed hypoglycemic events refer to all hypoglycemic events that had a glucose value ≤70 ml/dL or where assistance was required. Symptomatic hypoglycemic events were to be reported as adverse events. Investigator-defined hypoglycaemia adverse events include all events that investigator marked as 'Hypoglycaemic event' in CRFs, regardless of the reported term or blood glucose value. It may include hypoglycemia itself as reported term or any other symptoms that that investigator may have attributed to hypoglycemia (e.g. dizziness, hyperhidrosis, and asthenia).
Time Frame: During the course of the study (82 weeks)
Population: Treated set (TS). Treatment assignment as first medication taken.
Measure: Number; unit: participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 170 | 169 | 155
participants | 60 | 61 | 56

10. Secondary Outcome: The Occurrence of Treat to Target Efficacy Response, That is an HbA1c Under Treatment of <7.0% After 18, 54, and 78 Weeks of Treatment
Description: The occurrence of treat to target efficacy response, that is an HbA1c under treatment of <7.0% After 18, 54, and 78 weeks of treatment
Time Frame: Baseline, 18, 54 and 78 weeks
Population: FAS (NCF)
Measure: Number; unit: participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 165 | 167 | 154
participants
  18 weeks | 9 | 30 | 30
  54 weeks | 14 | 23 | 27
  78 weeks | 11 | 20 | 27
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Empagliflozin 10 mg vs Placebo at 18 weeks; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 4.096, 95% CI 2-sided [1.846 to 9.088]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Empagliflozin 25 mg vs Placebo at 18 weeks; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 4.636, 95% CI 2-sided [2.083 to 10.321]
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 10 mg; Empagliflozin 10 mg vs Placebo at 54 weeks; Test type: Superiority or Other; p = 0.1248, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 1.750, 95% CI 2-sided [0.856 to 3.575]
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Empagliflozin 25 mg vs Placebo at 54 weeks; Test type: Superiority or Other; p = 0.0132, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 2.423, 95% CI 2-sided [1.203 to 4.879]
Statistical Analysis 5: Comparison: Placebo vs Empagliflozin 10 mg; Empagliflozin 10 mg vs Placebo at 78 weeks; Test type: Superiority or Other; p = 0.0986, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 1.939, 95% CI 2-sided [0.884 to 4.256]
Statistical Analysis 6: Comparison: Placebo vs Empagliflozin 25 mg; Empagliflozin 25 mg vs Placebo at 78 weeks; Test type: Superiority or Other; p = 0.0024, Regression, Logistic; Logistic regression includes treatment, geographical region and baseline HbA1c; Odds Ratio (OR) = 3.239, 95% CI 2-sided [1.518 to 6.911]

ADVERSE EVENTS:
Time Frame: During the course of the study (82 weeks)
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Serious Adverse Events (participants affected / at risk) | 28/170 | 28/169 | 28/155
Other Adverse Events (participants affected / at risk) | 115/170 | 110/169 | 95/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=170) | Empagliflozin 10 mg (N=169) | Empagliflozin 25 mg (N=155)
Cystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 2 | 0
Coronary artery disease (Cardiac disorders) | 2 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Device failure (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0
Accident at home (Injury, poisoning and procedural complications) | 0 | 1 | 0
Accident at work (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Carotid endarterectomy (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=170) | Empagliflozin 10 mg (N=169) | Empagliflozin 25 mg (N=155)
Nasopharyngitis (Infections and infestations) | 22 | 20 | 17
Urinary tract infection (Infections and infestations) | 13 | 21 | 16
Upper respiratory tract infection (Infections and infestations) | 10 | 18 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 56 | 56 | 55
Hyperglycaemia (Metabolism and nutrition disorders) | 17 | 16 | 15
Depression (Psychiatric disorders) | 3 | 10 | 2
Dizziness (Nervous system disorders) | 12 | 18 | 7
Headache (Nervous system disorders) | 5 | 5 | 8
Hypertension (Vascular disorders) | 12 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 13 | 10 | 11
Nausea (Gastrointestinal disorders) | 12 | 9 | 8
Vomiting (Gastrointestinal disorders) | 5 | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 11 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 8
Fatigue (General disorders) | 2 | 10 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.